CLINICAL TRIAL: NCT01683487
Title: Delayed Antibiotic Treatment in Community-acquired Pneumococcal Pneumonia. Analysis of Risk Factors and Impact on the Outcome.
Brief Title: Delayed Antibiotic Treatment in Community-acquired Pneumococcal Pneumonia.
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: MM-CAP
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Observation — Observational study only, no intervention.

SUMMARY:
I. To investigate time measurement from emergency room admission to first antibiotic administration.

II. To evaluate risk factors for prolonged time to first antibiotic administration.

III. To correlate time measurement with Charlson comorbidity index and multimorbidity patterns.

IV. To investigate the impact of a delayed time to first antibiotic administration on the outcome

DETAILED DESCRIPTION:
In this retrospective cohort study, we plan to include all patients presenting with a community-acquired pneumococcal pneumonia at the University Hospital of Zurich between January 1, 2006 and June 30, 2012 (6½ years). The patients will be identified either with one or more blood culture pairs positive for S. pneumoniae or with a positive pneumococcal urine antigen assay in combination with the clinical diagnosis of CAP, which was based on the presence of select clinical features (e.g., cough, fever, sputum production, and pleuritic chest pain) and is supported by imaging of the lung, usually by chest radiography according to Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of CAP in adults [11].

CAP is not considered if the patient is discharged from a hospital less than 7 days before the current hospital admission, if the first blood culture or urinary antigen assay is obtained more than 1 week after hospital admission, or if the patient has no clinical diagnosis of CAP at the time of admission. Patients referred from or transferred to another hospital are excluded.

After identification of eligible patients upon microbiological results, medical records are reviewed using a standardized data collection questionnaire. Comorbidity is determined using the Charlson comorbidity index [10]. Additionally, all patients are classified according to the multimorbidity patterns proposed by Holden et al. [12]. These are:

1. arthritis, osteoporosis, other chronic pain, bladder problems, and irritable bowel;
2. asthma, chronic obstructive pulmonary disease, and allergies;
3. back/neck pain, migraine, other chronic pain, and arthritis;
4. high blood pressure, high cholesterol, obesity, diabetes, and fatigue;
5. cardiovascular disease, diabetes, fatigue, high blood pressure, high cholesterol, and arthritis; and
6. irritable bowel, ulcer, heartburn, and other chronic pain.

Time calculation is based upon the moment of emergency room (ER) admission.

ELIGIBILITY:
Inclusion criteria: Patients with community-acquired pneumococcal pneumonia, which was confirmed by

1. detection of Streptococcus pneumoniae in blood cultures, tracheal secretion or sputum OR/AND
2. positive urinary pneumococcal antigen AND
3. presence of cough and presence of one of the following signs/symptoms: new focal chest signs; dyspnoea; tachypnoea; fever AND
4. radiologic signs of pneumonia

Exclusion criteria: - Pneumonia of other cause (e.g. non-pneumococcal pneumonia)

* Hospital-acquired or ventilator-associated pneumonia
* Patients referred from or transferred to another hospital

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted and treated at the University Hospital of Zurich because of severe community-acquired pneumococcal pneumonia requiring hospilazation.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
In-hospital mortaliy | From day of admission until discharge or dead
  Mortality during hospitalization because of pneumococcal pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — University Hospital Zurich, Division of Internal Medicine
Locations (1):
- University Hospital Zurich, Division of Internal Medicine, Zurich, Canton of Zurich, Switzerland